CLINICAL TRIAL: NCT03486405
Title: A Randomized Control Trial: Returning to Run After Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kyle East, Major, United States Air Force, Keller Army Community Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KACH2018
Record Dates: First submitted 2018-02-07; First posted 2018-04-03 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study will be a randomized control trial crossover design.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will have no in person education by researchers. All education and running modification will be performed via video. Education on running form, a home exercise program, and a 4 week return to run program will be provided to the subjects through e-mail. They will also receive the same in person video analysis performed at weeks 0 (initial), 10 and 6 months to assess running kinematics.
  Interventions: Other: Intervention group
- Control group (Active Comparator): This group will have the same 4 week return to run program, home exercise program, and video analysis performed at weeks 0 (initial), 10 and 6 months to assess running kinematics.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — Control group runners will receive the same graduated return to run intervals and 4-week home exercise program. However, they will receive no video education during the initial 10 weeks.
  Arms: Control group
Other: Intervention group — Runners randomized to the intervention group will receive additional video tele-health instruction on how to transition to a non-rearfoot strike (NRFS) running pattern. Runners in the intervention group will have additional tele-health follow-ups at weeks 1, 2, 4,6, 8, and 10 using a tele-conferencing program and the Hudl Technique application. At each tele-health video follow-up participants will be emailed a questionnaire assessing their progress and function. At month 6 a final data collection session to include video analysis will be performed.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to examine the effectiveness of telehealth via video feedback to transition rear foot strike runners to non-heel strike runner following a lower extremity injury. Telehealth re-education gait training is much cheaper than in-clinic retraining sessions with a medical provider and could be much more widely used by both consumers and researchers as a training aid, a way to help alter running form, prevent running injuries and be used as a tool for use in the rehabilitation of running related injuries.

DETAILED DESCRIPTION:
A convenience sample of 30 runners from the United States Military Academy (USMA) at West Point, New York (NY) who are recovering from a lower-extremity injury and are interested in participating in a return to run program. Acceptable lower-extremity injuries can include stress fractures proximal to the ankle, anterior chronic exertional compartment syndrome (CECS), patella-femoral pain syndrome, osteoarthritis of the lower-extremity, iliotibial band syndrome, chronic lower-extremity pain and or any participant that may benefit from the following; shorter stride, increased step rate, reduced knee loading, and reduced ground reaction force average vertical loading rates (AVLR). All participants will be screened via questionnaire and physical assessment for inclusion / exclusion from the study. Upon enrollment runners will be randomized into two groups. Regardless of group, all runners will have their running form and foot strike pattern analyzed using an instrumented treadmill and high-speed motion capture initially and at week 10. Kinetic and kinematic data including AVLR, impulse, foot strike pattern (FSP), contact time, step length, and step rate will be recorded at these time points. Additionally, all runners will receive the same graduated return to run intervals and 4-week home exercise program. Runners randomized to the intervention group will receive additional video tele-health instruction on how to transition to a non-rearfoot strike (NRFS) running pattern. Runners in the intervention group will have additional tele-health follow-ups at weeks 1, 2, 4,6, 8, and 10 using a tele-conferencing program and the Hudl Technique application. At each tele-health video follow-up participants will be emailed a questionnaire assessing their progress and function. At month 6 a final data collection session to include video analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Pain free walking 2 miles in 35 minutes
2. Weight bearing dorsiflexion (WBDF) Range of Motion (ROM) 80% symmetry
3. 20 unassisted single leg heel raises
4. Recovering from a lower-extremity injury

Exclusion Criteria:

1. History of previous stress fracture / fracture of the foot
2. Participant who already uses a non-rearfoot strike running pattern
3. Participant is pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Foot Strike Pattern | 6 months
  Analyzed through slow motion camera on an instrumented treadmill.

SECONDARY OUTCOMES:
Perceived running pain | 6 months
  Subjects will self evaluate running ease and efficiency through the Single Assessment Numeric Evaluation.
Perceived running effort | 6 months
  Subjects will self evaluate running ease and efficiency through the University of Wisconsin Running Injury and Recovery Index.
Perceived effort of running | 6 months
  Subjects will self evaluate running ease and efficiency through the Patient Specific Functional Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No
The principal investigator will keep your research records. These records may be looked at by staff from the Keller Army Community Hospital Department of Clinical Investigation, the Keller Army Community Hospital (KACH) Institutional Review Board (IRB), the Army Clinical Investigation Regulatory Office (CIRO), the Department of Defense (DoD) Higher Level Review, and other government agencies as part of their duties.
  These duties include making sure that the research participants are protected. Your research records may be disclosed outside of the hospital, but in this case, you will be identified only by a unique code number. Information about the code will be kept in a secure location and access limited to authorized research study personnel.
  This research study meets the confidentiality requirements of the Health Insurance Portability and Accountability Act (HIPAA).